CLINICAL TRIAL: NCT03730792
Title: SHIFT Onboard: Protecting New Transit Operators Against Safety and Health Hazards
Brief Title: Success & Health Impacts For Transit Drivers During Onboarding
Acronym: SHIFT Onboard
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ryan Olson, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20047; 2R01HL105495-06A1 (NIH)
Record Dates: First submitted 2018-10-30; First posted 2018-11-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: Body Weight; Nutrition; Physical Activity; Sleep; Stress; Occupational Health; Working Conditions
MeSH Terms: conditions — Obesity; Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHIFT Onboard Intervention (Experimental): A 12-month onboarding process and social challenge supported with goal setting, computer-based training, self-monitoring, and group motivational interviewing.
  Interventions: Behavioral: SHIFT Onboard Intervention
- Usual Practice Control (No Intervention): Participants experience standard or "Usual Practices" in new employee onboarding processes at their workplace.

INTERVENTIONS:
Behavioral: SHIFT Onboard Intervention — A 12-month onboarding process and social challenge supported with goal setting, computer-based training, self-monitoring, and group motivational interviewing.
  Arms: SHIFT Onboard Intervention

SUMMARY:
The project is a cluster randomized controlled trial of an occupational health intervention for newly hired bus operators. Transit authorities will be randomized to intervention and usual practice conditions and new bus operators will be recruited to participate in a two year study. Intervention participants will complete a program designed to prevent weight gain while also supporting early adjustment and job success. Control participants will experience standard or usual practice working conditions.

DETAILED DESCRIPTION:
Epidemiological evidence indicates that bus driving is associated with increased risk for obesity and some chronic diseases, and that it is time for interventions. In this regard, the early transition into bus driving has been neglected. Not only are interventions lacking for new employees entering potentially obesogenic occupations, but workplace training and socialization programs for new hires (referred to as onboarding) rarely address potential occupational health hazards.

To address research gaps, investigators will integrate an effective health intervention approach with traditional onboarding programs for new bus drivers. This intervention approach, which was originally developed with commercial truck drivers, was implemented through a mobile friendly website, and tactics included an incentivized game-like competition that was supported with behavior and body weight logging, computer-based training, and motivational interviewing. In a cluster-randomized trial with commercial truck drivers the intervention produced a mean body weight effect of -7.29 lbs (p<.0001; Olson et al, 2016), which is among the strongest results observed globally with occupational drivers.

In the proposed intervention adaptation, the "SHIFT Onboard" intervention (Success & Health Impacts For Transit drivers during Onboarding) will be designed to prevent weight gain among new bus drivers while also supporting early adjustment and job success. The primary hypotheses are that relative to usual practice, SHIFT Onboard participants will have (1) superior energy balance behaviors (sleep, eating, exercise) and (2) less weight gain. Investigators will also evaluate impacts on new employee adjustment and economic outcomes that are critical to employers; the ultimate adopters of occupational health interventions. This project will take place over five years and will accomplish three specific aims:

1. Adapt proven tactics and pilot SHIFT Onboard with new bus drivers: Through formative research with transit partners and iterative testing with drivers investigators will adapt existing web technology, intervention tactics, and training content for newly hired mass transit bus drivers. The adapted SHIFT Onboard intervention will then be pilot tested with new drivers at a partner transit authority.
2. Determine the efficacy of SHIFT Onboard for preventing weight gain. Metropolitan transit authorities, stratified by size, will be randomly assigned to intervention or usual practice control conditions. SHIFT Onboard will be implemented with natural groups of bus operators who complete training together during the first year. Primary intervention effectiveness outcomes will be between-groups differences at 1- and 2-year follow-ups in changes in energy balance behaviors (sleep, eating, exercise) and body weight.
3. Evaluate new employee adjustment and economic impacts of SHIFT Onboard. Investigators will also evaluate intervention impacts on new bus operator adjustment (role stress, confidence, connectedness) and job attitudes (job satisfaction, intention to remain). Economic return on investment calculations will contrast intervention costs relative to savings projected from intervention effects (e.g., health care costs, absenteeism, safety).

Investigators will also collect measures of work demands, stressors, and strains (responses to stressors) at all time points to characterize occupational exposures among the sample, and to explore for possible associations with workers' health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hired to work as a transit bus operator at a participating transit authority, and currently in the pre-service training period

Exclusion Criteria:

* Female participants who are pregnant or become pregnant during the study period will be excluded from body weight related intervention activities and outcome analyses

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2020-03-22 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body weight at 12 and 24 months | Baseline, 12, and 24 months
  Directly measured body weight in kg.
Body Mass Index | Baseline, 12 and 24 months
  Calculated from directly measured weight and height (kg/m^2).
Change from baseline in percent body fat | Baseline, 12 and 24 months
  Percent body fat measured through bioelectric impedence
Change from baseline in self-reported fruit and vegetable intake at 12 and 24 months | Baseline, 12, and 24 months
  Survey measures of fruit and vegetable intake.
Change from baseline in self-reported consumption of high fat foods at 12 and 24 months. | Baseline, 12 and 24 months.
  Survey measure of high fat food consumption frequency and portion sizes.
Change from baseline in self-reported sugary food and drink consumption at 12 and 24 months | Baseline, 12 and 24 months.
  Survey measure of the frequency of sugary food and drink consumption.
Change from baseline in self-reported fast food consumption. | Baseline, 12 and 24 months.
  Survey measure of the frequency of fast food consumption.
Change from baseline in self-reported physical activity at 12 and 24 months | Baseline, 12, and 24 months
  Survey measures of daily/weekly physical activity levels.
Change from baseline in actigraphically measured physical activity at 12 and 24 months | Baseline, 12 and 24 months
  Actigraphy measures of daily/weekly of physical activity levels.
Change from baseline in self-reported sleep quality at 12 and 24 months | Baseline, 12, and 24 months
  Survey measures of typical sleep quality.
Change from baseline in self-reported sleep quantity at 12 and 24 months | Baseline, 12 and 24 months
  Survey measures of typical daily sleep time.
Change from baseline in actigraphically measured sleep quality at 12 and 24 months | Baseline, 12 and 24 months
  Actigraphy measures of sleep quality as indicated by minutes of Wake After Sleep Onset in main sleep periods.
Change from baseline in actigraphically measured sleep quantity at 12 and 24 months | Baseline, 12 and 24 months
  Actigraphy measures of sleep duration in minutes for the daily main sleep period and naps.

SECONDARY OUTCOMES:
Changes in job role conflict | Baseline, 12, and 24 months
  Survey measures of job role conflict.
Changes in perceived acceptance by others | Baseline, 12 and 24 months
  Survey measures of perceived acceptance by others.
Changes in job-related self-efficacy | Baseline, 12 and 24 months
  Survey measures of job-related self-efficacy.
Changes in job satisfaction | Baseline, 12 and 24 months
  Survey measure of job satisfaction
Changes in intention to remain at job | Baseline, 12 and 24 months
  Survey measures of intention to remain.
Economic cost-benefit factors | 12 month intervention costs, and a target minimum of four years of corporate data for each agency (2 historical, 2 during study period)
  Intervention costs (e.g., participant wages, fees for group facilitators, cost of resources/tech support, intervention incentives) will be contrasted with estimated savings (e.g., estimates of health care cost savings based on weight changes, and estimates of costs/savings utilizing corporate data for study participants on absenteeism, job turnover, bus collisions, driver injuries and workers' compensation claims, and passenger/pedestrian/other driver injuries).
Absenteeism | Baseline, 12 and 24 months
  Organizational records of absenteeism for new bus operators
Job turnover | Baseline, 12 and 24 months
  Organizational records of job turnover among new bus operators
Bus collisions | Baseline, 12 and 24 months
  Organizational records of bus collisions among new bus operators
Injuries | Baseline, 12 and 24 months
  Organizational records of bus operator and passenger injuries

OTHER OUTCOMES:
Baseline body weight as a moderator of intervention effects on weight at follow-ups | Baseline, 12, and 24 months
  Baseline body weight evaluated as a moderator of intervention effects at 12 and 24 months.
Change from baseline in blood pressure at 12 and 24 months | Baseline, 12, and 24 months
  Direct measurement in mmHg.
Change from baseline in triglycerides | Baseline, 12, and 24 months
  Direct measurement of triglycerides via Cholestech LDX Analyzer in mg/dL.
Change from baseline in Hemoglobin A1c at 12 and 24 months | Baseline, 12, and 24 months
  HbA1c measured via fingerprick blood sample.
Change from baseline in Total cholesterol | Baseline, 12, and 24 months
  Total cholesterol measured from fingerstick blood sample via Cholestech LDX Analyzer in mg/dL.
Change from baseline in HDL cholesterol | Baseline, 12 and 24 months
  HDL measured from fingerstick blood sample via Cholestech LDX Analyzer in mg/dL.
Change from baseline in LDL cholesterol | Baseline, 12 and 24 months
  LDL measured from fingerstick blood sample via Cholestech LDX Analyzer in mg/dL.
Change from baseline in the LDL/HDL cholesterol ratio | Baseline, 12, and 24 months
  LDL/HDL cholesterol ratio computed from values measured via Cholestech LDX Analyzer in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Olson, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson R, Wipfli B, Thompson SV, Elliot DL, Anger WK, Bodner T, Hammer LB, Perrin NA. Weight Control Intervention for Truck Drivers: The SHIFT Randomized Controlled Trial, United States. Am J Public Health. 2016 Sep;106(9):1698-706. doi: 10.2105/AJPH.2016.303262. Epub 2016 Jul 27. PMID 27463067